CLINICAL TRIAL: NCT05006443
Title: Staging Classification of Severe Tricuspid Regurgitation Using Novel Cardiac Imaging Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mohamad Adnan Alkhouli, Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-003928
Record Dates: First submitted 2021-07-31; First posted 2021-08-16 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moderate or severe tricuspid regurgitation (Other): 40 patients with moderate or more TR on echocardiography will undergo CMR/MRE with contrast to assess TR severity, and the associated extra-valvular cardiac and liver abnormalities. Patients will continue their clinical management by their primary physicians as per the standards of care. 1-year follow up will be conducted via phone to inquire about patient's vital status (dead/alive), symptoms and hospitalizations.
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance — a non-invasive assessment to determine severity of tricuspid regurgitation
  Other Names: Cardiac MRI

SUMMARY:
The purpose of this research is to assess the severity of tricuspid regurgitation (a disorder in which the tricuspid valve in the heart does not close tight enough) using cardiac magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
40 patients with moderate or more TR on echocardiography will undergo CMR/MRE with contrast to assess TR severity, and the associated extra-valvular cardiac and liver abnormalities as shown in the flow diagram below. Patients will continue their clinical management by their primary physicians as per the standards of care. 1-year follow up will be conducted via phone to inquire about patient's vital status (dead/alive), symptoms and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or more tricuspid regurgitation

Exclusion Criteria:

1. Prior tricuspid valve prosthesis
2. Pacemaker/defibrillator that would impede MRI imaging
3. Planned tricuspid valve surgery
4. Primary liver pathology

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Severity of tricuspid regurgitation by cardiac magnetic resonance imaging | 1 year
  Incidence of severity of TR by CMR as compared with current gold standard (TTE)

SECONDARY OUTCOMES:
Correlation between severity of Tricuspid regurgitation by cardiac magnetic resonance imaging vs. elastography | 1 year
  Correlation between severity of TR by CMR vs. echocardiography with 1-year composite endpoint of death, heart failure hospitalization, or tricuspid valve surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Alkhouli, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials